CLINICAL TRIAL: NCT03295448
Title: Circulating Fatty Acids as Biomarkers of Dietary Carbohydrates: a Randomized Trial
Brief Title: Fatty Acid Biomarkers of Carbohydrate Intake
Acronym: CARBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CARBIO
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Dyslipidemias
Keywords: fatty acids; biomarker; carbohydrate; lipogenesis
MeSH Terms: conditions — Dyslipidemias | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Fat - Sugar - Fiber (Active Comparator): Intervention: consuming diets rich in fat, rich in sugar, and rich in fibers during treatment periods 1, 2, and 3, respectively. Treatment periods are separated by one week of habitual diet.
  Interventions: Other: Low carbohydrate diet; Other: High carbohydrate, high sugar diet; Other: High carbohydrate, low sugar diet
- Fat - Fiber - Sugar (Active Comparator): Intervention: consuming diets rich in fat, rich in fiber, and rich sugar during treatment periods 1, 2, and 3, respectively. Treatment periods are separated by one week of habitual diet.
  Interventions: Other: Low carbohydrate diet; Other: High carbohydrate, high sugar diet; Other: High carbohydrate, low sugar diet
- Sugar - Fiber - Fat (Active Comparator): Intervention: Consuming diets rich in sugar, rich in fiber, and rich in fat during treatment periods 1, 2, and 3, respectively. Treatment periods are separated by one week of habitual diet.
  Interventions: Other: Low carbohydrate diet; Other: High carbohydrate, high sugar diet; Other: High carbohydrate, low sugar diet
- Sugar - Fat - Fiber (Active Comparator): Intervention: Consuming diets rich in sugar, rich in fat, and rich in fiber during treatment periods 1, 2, and 3, respectively. Treatment periods are separated by one week of habitual diet.
  Interventions: Other: Low carbohydrate diet; Other: High carbohydrate, high sugar diet; Other: High carbohydrate, low sugar diet
- Fiber - Sugar - Fat (Active Comparator): Intervention: Consuming diets rich in fiber, rich in sugar, and rich in fat during treatment periods 1, 2, and 3, respectively. Treatment periods are separated by one week of habitual diet.
  Interventions: Other: Low carbohydrate diet; Other: High carbohydrate, high sugar diet; Other: High carbohydrate, low sugar diet
- Fiber - Fat - Sugar (Active Comparator): Intervention: consuming diets rich in fiber, rich in fat, and rich in fiber during treatment periods 1, 2, and 3, respectively. Treatment periods are separated by one week of habitual diet.
  Interventions: Other: Low carbohydrate diet; Other: High carbohydrate, high sugar diet; Other: High carbohydrate, low sugar diet

INTERVENTIONS:
Other: Low carbohydrate diet — Diet low in carbohydrates (38%E), but higher in total and saturated fat.
Other: High carbohydrate, high sugar diet — Diet high in carbohydrates (53%E) and sugars, but low in wholegrain, rye and wheat fibre.
Other: High carbohydrate, low sugar diet — Diet high in carbohydrates (53%E), wholegrain, rye and wheat fibre, but low in sugars.

SUMMARY:
The overall aim is to investigate if circulating fatty acids and lipids are influenced by alterations in carbohydrate amount and quality.

DETAILED DESCRIPTION:
In this isocaloric clinical cross-over trial, the investigators aim to investigate if circulating fatty acids and lipids are influenced by alterations in carbohydrate amount and quality. The investigators intend to evaluate if changes in carbohydrate quantity and quality (including sugar) influence circulating even-chain saturated fatty acids or if fatty acid-derived indices of desaturation and de novo lipogenesis are more sensitive biomarkers of carbohydrate intake. By performing untargeted lipidomic analyses, the investigators aim to search for novel lipid biomarkers of carbohydrate quantity and quality. The investigators also want to evaluate the influence of moderate alterations of carbohydrate and sugar intake on lipoproteins, insulin sensitivity, inflammatory proteins.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-38

Exclusion Criteria:

* abnormal lab tests (assessed by screening and judged by a physician), diabetes, cardiovascular, kidney, liver or malignant disease, and weight-loss (±3kg) the preceding 3 months of screening. Extreme diets, i.e. very-low carbohydrate diets, intermittent fasting, vegan diets or allergic to gluten

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Palmitic acid in different plasma fractions | 14-20 days
  Measured by liquid gas chromatography (GC)

SECONDARY OUTCOMES:
Even-chain saturated fatty acids (i.e. 14:0, 18:0) and monounsaturated fatty acids | 14-20 days
  Measured by liquid GC

OTHER OUTCOMES:
Desaturation indices end lipogenic indices | 14-20 days
  These indices are product-to-precursor fatty acids measured by GC

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Riserus, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala univeristy hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Bajahzer MF, Rosqvist F, Friden M, Iggman D, Pingel R, Marklund M, Riserus U. Contrasting Carbohydrate Quantity and Quality and the Effects on Plasma Saturated and Monounsaturated Fatty Acids in Healthy Adults: A Randomized Controlled Trial. J Nutr. 2023 Mar;153(3):683-690. doi: 10.1016/j.tjnut.2023.01.005. Epub 2023 Jan 13. PMID 36797136